CLINICAL TRIAL: NCT02484937
Title: Improving Functional Outcomes and Lowering Health Care Costs by Enhanced Integration of Primary Care Providers and Pain Medicine Physicians for Chronic Non-cancer Pain Patients
Brief Title: Improving Outcomes and Lowering Costs by Integration of Primary Care Providers and Pain Medicine Physicians for Pain Pts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Rush University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Asokumar Buvanendran, Professor, Department of Anesthesiology, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14100602
Record Dates: First submitted 2015-06-19; First posted 2015-06-30 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Back Pain; Chronic Pain; Pain, Intractable
Keywords: Pain management
MeSH Terms: conditions — Back Pain; Chronic Pain; Pain, Intractable; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (PMS Treatment) (Active Comparator): Subjects will be treated monthly for 6 months by Pain Medicine Specialist (PMS) per standard protocol. The PCP will not be involved in the treatment.
  Interventions: Other: Group 1 (PMS Treatment)
- Group 2 (PCP Treatment) (Experimental): Subjects will be treated monthly for 6 months by the Primary Care Provider (PCP).The PCP will be involved and a multimodal therapeutic strategy will be communicated to the PCP by the PMS. The PCP will make dosage based on an algorithm provided by the PMS on how to adjust drug doses over time. It is not intended that the PCP may have ongoing engagement with the PMS. A direct line of communication will be set up between the PCP and the data integration clinical coordinator to handle serious medical concerns.
  Interventions: Other: Group 2 (PCP Treatment)

INTERVENTIONS:
Other: Group 2 (PCP Treatment) — For the PCP group treatment will be performed (pain treatment/medications) by the Primary Care Physician in his/her office/clinic.
  Arms: Group 2 (PCP Treatment)
Other: Group 1 (PMS Treatment) — For the PMS group treatment will be performed (pain treatment/medications) by the Pain Medicine Specialist in his/her office/clinic.
  Arms: Group 1 (PMS Treatment)

SUMMARY:
This study will demonstrate that functional improvement measures over a 6-month period for chronic low back patients under the care of Primary Care Provider (PCP), using a therapeutic plan formulated initially by the Pain Medicine Specialist (PMS), are equivalent to those under the care of the PMS only. Chronic low back pain patient will be initially be evaluated by the PMS. If no interventional pain therapy is required, a multimodal therapeutic plan (pharmacological and/or non-pharmacological) will be formulated to manage the chronic low back pain. Patients will be randomized into one of the two groups: Group 1 - Subjects will be treated monthly for the following 6 months by PMS, and Group 2 - Subjects will be treated by their own PCP for monthly visits for 6 months.

DETAILED DESCRIPTION:
In this trial, each chronic low back pain patient presenting to the Rush University Pain Center will initially be evaluated by the PMS.The initial evaluation visit, as part of the routine care for all new low back patients, will include the following: a full physical examination, review of medical health and medication history, and radiological imaging (EHR will be used for the study). In addition, all new patients will need to provide a urine drug screening test and will need to undergo psychological testing and evaluation.

A determination will be made by the PMS on whether the best treatment modality includes an interventional approach or non-interventional. If no interventional pain therapy is required, a multimodal therapeutic plan (pharmacological and/or non-pharmacological) will be formulated to manage the chronic low back pain. A complete workup will be performed to accomplish this task.

If a non-interventional treatment (pharmacological and non-pharmacological) is selected, that can be implemented by a PCP, the patients will be informed of the study, and if interested, a Prescreening Informed Consent and Health Insurance Portability and Accountability Act (HIPAA) form will be obtained from patient to give permission to contact their PCP. At that point, the patients' PCPs will be contacted, presented with the study information, and asked if they want to participate in the study. If the PCP agrees, the Main Study Informed Consent will be obtained from the patient. Patients meeting criteria would then be randomized into one of two treatment groups for continued treatment over the next 6 months. This initial multimodal therapeutic treatment can be altered by the respective treatment groups (PMS or PCP) to which study subject has been randomized.

Group 1 (PMS treatment): Subjects will continue to be followed for the next 6 months by the PMS (typically every month for the treatment of chronic pain) per standard protocol. The PCP will not be involved in the treatment.

Group 2 (PCP treatment): Subjects will be followed by the PCP for the next 6 months. The PCP will be involved using EHR and a multimodal therapeutic strategy will be communicated to the PCP by the PMS. The PCP will make dosage based on an algorithm provided by the PMS on how to adjust drug doses over time (general template-See below). It is not intended that the PCP may have ongoing engagement with the PMS. While the PCP may request clarification by the PMS during the first week of subject treatment, any further contact between the PCP and the PMS would result in the subjects being withdrawn from the study. In addition, a direct line of communication will be set up between the PCP and the data integration clinical coordinator to handle serious medical concerns. In case of serious medical events, the subject will be withdrawn from the study and appropriate medical care will be provided by the PMS or PCP.

Group 1 & 2: Subjects in both groups will undergo the following:

1. Urine drug screening test (qualitative); includes amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, ethanol, and opioids
2. Receive a sample copy of an opioid contract/agreement
3. PMS will query the Illinois prescription monitoring program for that patient to determine the various health care providers who are prescribing narcotics or other controlled medications.
4. Undergo a psychological test and evaluation by the Rush University Pain Center psychologist (including the Screener and Opioid Assessment for Patients with Pain-Revised (SOAPP-R)13), to determine risk of drug abuse.

Template for treatment of low back pain to be provided for PCP.

This template is only a suggestion, and clinical and medical judgment for each patient will be decided by the PMS. Listed are the categories of pharmacological and non-pharmacological modalities, but the PMS will formulate a patient-specific prescriptive plan after evaluation at the initial work-up:

1. Non-steroidal anti-inflammatory drugs (NSAIDs): preferably COX-2 inhibitor for all patients. If NSAIDs are prescribed, GI prophylaxis needs to be provided.14,15 This would be prescribed to all patients and will be provided daily and not 'as needed' medication, unless there are adverse events that prevent its administration.
2. Muscle relaxants: such pharmacological agents include baclofen, tizanidine, or lorazepam to relieve painful muscle spasms16
3. Opioids: long-acting opioids (oxycodone, controlled- release), short-acting opioids (e.g. hydrocodone/acetaminophen)14,15,17
4. Anticonvulsants: mainly gabapentin or pregabalin18
5. Transcutaneous electrical nerve stimulation (TENS) unit19 At the end of the 6-month treatment period (end of study), patients will be given the option to continue the treatment with their group or changing to any other treatment available.

A research study nurse, blinded to group allocation, will call patients (from both groups) every month to collect BPI questionnaire responses over the phone. In addition, a general measure of functional health and well-being, the SF-36 health-related quality of life outcome measure (Short-Form 36 Health Survey), will be collected during the same call.21 The SF-36 total score can be used as an overall health measure, or as a measure of two different health domains: physical health (including bodily pain) and mental health, as well as further division into more specific subscales. A baseline BPI and SF-36 will be obtained from each subject's initial visit record (EHR). The research study nurse will enter data obtained from the phone calls directly into the Rush University Pain Centers (RUPC) EHR on the eClinicalWorks platform.

To evaluate procedural variations, side effects and secondary outcomes over the 6 month follow-up treatment period, a data integration clinical coordinator (DICC), not blinded to group allocation, will query electronic and physical health records, from both the PCP and PMS, as well as corresponding HIS's.

ELIGIBILITY:
Inclusion Criteria:

1.Non-structural non-specific chronic low back pain of a least 3 months duration

2.18 years of age or older

3.Has a primary care provider (PCP)

Exclusion Criteria:

1. Unable to communicate with health care providers
2. Refuses to complete the required outcome measures
3. Unable to provide consent
4. Advanced medical illness (severe systemic disease)
5. Significant psychiatric history: a diagnosis of schizophrenia, bipolar disorder, or severe depression.
6. History of psychosis or psychiatric hospitalization, suicidal ideation or attempt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Pain interference with daily activity - BPI score change from baseline. | 6 months
  The Brief Pain Inventory (BPI) short form is a self-report questionnaire using items (questions) on a 11-point scale (0-10), and will be used to assess impact of pain on daily activities, and pain severity.
  We will gather data approximately on a monthly basis (Baseline, 1 month, 2 month, 3 month, 4 month, 5 month, 6 month).

SECONDARY OUTCOMES:
Procedural variations | 6 months
  A data integration clinical coordinator (DICC), not blinded to group allocation, will query electronic and physical health records, from both the PCP and PMS
Functional health and well-being - improvement from baseline | 6 months
  The Short Form-36 Health Survey (SF-36) form is a health-related quality of lif questionnaire which measures two different health domains: physical health (including bodily pain) and mental health, as well as further division into more specific subscales.
Patients experience of care | 6 months
  The Patient Satisfaction Questionnaire (PSQ-18) assesses global satisfaction with medical care as well as satisfaction with six aspects of care: technical quality, interpersonal manner, communication, financial aspects of care, time spent with doctor, and accessibility of care

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States